CLINICAL TRIAL: NCT04908735
Title: Ruxolitinib for Early Lung Dysfunction After HSCT: a Phase II Study
Brief Title: Ruxolitinib for Early Lung Dysfunction After Hematopoietic Stem Cell Transplant
Acronym: HSCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0719
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic Stem Cell Transplant (HSCT); Bronchiolitis Obliterans (BO)
MeSH Terms: conditions — Bronchiolitis Obliterans | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib Treatment (Experimental)
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Participants will receive ruxolitinib orally twice daily for 24 weeks.

SUMMARY:
Hematopoietic stem cell transplant (HSCT) is an effective but toxic therapy, and lung injury affects as many as 25% of children receiving HSCT. Improved transplant techniques and major improvements in survival mean that HSCT is being more widely used, and more mismatched grafts are being used. Bronchiolitis obliterans (BO) is a major limitation of pediatric HSCT success as BO is commonly diagnosed late in children, when lung injury is irreversible, leading to long term morbidity or even death. Currently, there are major gaps in our knowledge regarding incidence, etiology and optimal treatment of BO following HSCT, and important diagnostic limitations specific to children. Diagnosis of BO is usually based on performance of pulmonary function tests, which is usually impossible in ill children under 10. Even older children who feel unwell or un-cooperative may be unable to produce interpretable data. These deficiencies in diagnosis mean that BO is commonly diagnosed late, meaning fibrosis has occurred and lesions are irreversible.

The hypothesis for this interventional trial is that early treatment with standard Flovent/montelukast and steroids plus ruxolitinib will reverse lung injury and reduce the frequency of chronic pulmonary impairment or florid BO.

ELIGIBILITY:
Inclusion Criteria:

Subjects ≥ 5 years and ≤ 60 years of age who have undergone allogeneic HCT AND exhibit early lung dysfunction as defined by any one of the following:

* >10% decrease in FEV1 from baseline or decrease of 25% of FEF 25-75 from baseline
* active GVHD in another organ system + pulmonary symptoms (Tachypnea without wheezing, new oxygen requirement, cough)
* Increased R5 by 50% by clinical oscillometry
* Air trapping on CT, small airway thickening, or bronchiectasis

AND - All age groups, including adults:

Adequate renal function defined as estimated Creatinine Clearance (CrCl) ≥ 30 mL/min as calculated by the cystatin c GFR or nuclear GFR

Adequate hepatic function as defined by:

* ALT and AST ≤ 5 x ULN, unless the ALT / AST increase is due to cGVHD
* Total bilirubin of ≤ 5 x ULN (unless of non-hepatic origin or due to Gilbert's Syndrome) or Total bilirubin of < 10 x ULN if due to GVHD

Adequate hematological function defined as:

* Absolute neutrophil count ≥1.0 x 10^9/L
* Platelets ≥30 x 10^9/L

PT/INR <2 x ULN and PTT (aPTT) < 2 x ULN (unless abnormalities are unrelated to coagulopathy or bleeding disorder)

Exclusion Criteria:

* Known hypersensitivity to any constituent of the study medication.
* Active uncontrolled pulmonary infection (preceding infectious evaluation including bronchoscopy as clinically indicated)
* Subjects who are pregnant or breastfeeding or are at risk of pregnancy or fathering a baby and are unable to use acceptable highly effective method of birth control (e.g., implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete abstinence or sterilized partner) and a barrier method (e.g., condoms, cervical ring, sponge, etc.) during the period of therapy and for 90 days for both females and males after the last dose of study drug.
* Subjects previously treated with investigational agent for GVHD within the 30 days prior to first dose of study treatment. Other non-GVHD additional investigational agents may be allowed on a case by case basis with review/approval by the study Lead PI.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with ruxolitinib treatment response | 6 months from early lung dysfunction diagnosis
  Treatment response is defined by stable and/or improved lung function as defined by the National Institutes of Health Chronic GVHD Response Criteria Working Group.

SECONDARY OUTCOMES:
Percentage of participants with JAK inhibition | 24 weeks after ruxolitinib initiation
  The presence of JAK inhibition will be measured by phospho stat5
Number of participants with lung function response measured by a Xenon MRI scan | 24 weeks after ruxolitinib initiation
  The presence of a lung function response will be measured by a Xenon MRI scan
Number of participants with lung function response measured by oscillometry | 24 weeks after ruxolitinib initiation
  The presence of a lung function response will be measured by oscillometry
Number of participants with lung function response measured by home spirometry | 24 weeks after ruxolitinib initiation
  The presence of a lung function response will be measured by home spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Kasiani Myers, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - University of Minnesota, Minneapolis, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania